CLINICAL TRIAL: NCT04431999
Title: Evaluation of a Transfusion Therapy Using Whole Blood Versus Fractionated Blood Products in the Management of Coagulopathy in Patients Admitted to Hospital for Acute Traumatic Hemorrhage
Brief Title: Evaluation of a Transfusion Therapy Using Whole Blood in the Management of Coagulopathy in Patients With Acute Traumatic Hemorrhage
Acronym: T-STORHM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Collaborators: TIMC-IMAG (Other); Floralis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A02706-51
Record Dates: First submitted 2020-05-28; First posted 2020-06-16 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-02

CONDITIONS: Trauma; Acute Hemorrhage; Coagulopathy
Keywords: Whole Blood; Acute traumatic coagulopathy; Transfusion
MeSH Terms: conditions — Wounds and Injuries; Hemostatic Disorders | interventions — Exchange Transfusion, Whole Blood

STUDY DESIGN:
Intervention Model Description: Multicenter, Controlled, Randomized, Open Labe Therapeutic Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole blood group (Experimental): Damage control resuscitation for trauma care using whole blood.
  Interventions: Drug: Whole blood transfusion
- Fractionated blood products group (Active Comparator): Damage control resuscitation for trauma care using component therapy.
  Interventions: Drug: Fractionated blood products transfusion

INTERVENTIONS:
Drug: Whole blood transfusion — Severe trauma patients with a life threatening bleeding will be managed with 3 whole blood bags for the 1st and 2nd pack. The later packs will consist of 3 packed red blood cells (PRBCs), 3 plasma units and 1 dose of platelets.
  Arms: Whole blood group
Drug: Fractionated blood products transfusion — Severe trauma patients with a life threatening bleeding will be managed with 3 packed red blood cells (PRBCs), 3 lyophilised plasma units and 1 dose of platelets for the 1st. The 2nd pack will consist of 3 packed red blood cells (PRBCs) and 3 lyophilised plasma units. Then, the later pack will consist of 3 packed red blood cells (PRBCs), 3 plasma units and 1 dose of platelets.
  Arms: Fractionated blood products group

SUMMARY:
The prognosis of traumatized hemorrhages is correlated with the nature of transfusion therapy: a 50% reduction in mortality for an early and massive supply of plasma, and 20% for an early and massive supply of platelets. However, this strategy encounters logistical difficulties, particularly in a context of collective emergency (attacks). The use of whole blood, widely documented by the Armed Forces, improves the availability of plasma and platelets, and simplifies handling by the various actors in the chain.

T-STORHM is a randomized, controlled, parallel clinical trial.This study tests non-inferiority of whole blood transfusion therapy in the management of coagulopathy in patients with acute traumatic hemorrhage.

DETAILED DESCRIPTION:
In recent years, terrorist attacks have confronted the investigator's healthcare system with a massive influx of victims of war weapon injuries. This new fact makes the efficiency of transfusion therapy crucial: hemorrhage is the leading cause of death from weapons of war, and the high number of victims of each attack changes the logistical approach.

The logistical problems with transfusion therapy, including red blood cell (PRBCs), plasma and platelet concentrates, are the speed of delivery and availability. Using whole blood is a pragmatic solution to overcome these problems. This solution has been used for many years by the French Army to ensure platelet transfusion in traumatic hemorrhages

The hypothesis of the T-STORHM study is that the use of whole blood is a solution in a context of civil trauma not effective less than component therapy (PRBCs, plasma and platelet concentrates) in the management of coagulopathy in patients admitted to hospital for traumatic hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

Severe trauma patients requiring the initiation of a massive transfusion protocol determined on

1. At least two Red flag score factors (according to pre-hospital data) :

   * Suspected pelvic fracture
   * Shock index (FC / PAS)> = 1
   * Microdose hemoglobin <13g
   * Average blood pressure <70 mmHg
   * Need for prehospital tracheal intubation
2. AND at least two criteria of the Assessment of Blood Consumption (ABC) score established at the patient's arrival:

   * Penetrating trauma
   * Focused Abdominal Sonography for Trauma (FAST) echo positive
   * Blood pressure <90 mmHg
   * Respiratory rate >120 bpm
3. AND/OR after clinical assessment and on the prediction of the practitioner in charge of the treatment of the injured person of the need to transfuse during the emergency management of the injured person

Exclusion Criteria:

* Non-traumatic hemorrhage
* Patients transfused with more than two PRBCs before the initiation of the massive transfusion protocol.
* Anti-coagulation treatment
* Pregnancy
* Age < 18 years
* Patient refusing administration of blood products
* Patient transferred from another hospital
* Patient nor transported by a physician-staffed prehospital emergency medical system
* Burn patient (≥30% of body surface).
* Patient under specific known transfusion protocol (for example : allo immunization...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-12-04 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Non inferiority on the correction of coagulopathy, during emergency transfusion of bleeding trauma using whole blood compared to the use of component therapy (packed red blood cells, plasma units and platelets). | 6 hours following hospital admission
  This outcome is measured on the correction of traumatic coagulopathy, measured by the value of a viscoelastometric parameter : the maximum amplitude (MA) (measured by a thromboelastogram).

SECONDARY OUTCOMES:
Effectiveness of circulatory resuscitation | 2 hours following hospital admission
  Proportion of patients with lactate clearance > 20% per hour at H2.
Mortality | 2 hours following hospital admission and Day 30 (or the last day of hospitalization)
  Number of deaths.
Mortality / Morbidity | 24 hours following hospital admission
  Composite endpoint : Number of deaths at H24 or impairment of vital functions with a Sequential Organ Failure Assessment (SOFA) score greater than or equal to 12.
Impact on timeframe to obtain blood products | 2 and 6 hours following hospital admission
  Time to obtain product ratios in accordance with recommendations.
Impact on time to start transfusion therapy | Time between admission and transfusion therapy
  Time to start transfusion therapy.
Evolution of coagulopathy. | At inclusion, 2, 6 and 24 hours following hospital admission
  All the parameters of the thrombelastography (TEG) (R/CK, alpha/CK, MA/CRT, LY30/CK, MA/CFF and TEG-ACT/CRT) allow to evaluate the coagulopathy.
Evolution of coagulopathy | At inclusion, 2, 6 and 24 hours following hospital admission.
  All the parameters of the coagulation (PT, APTT, fibrinogene) allow to evaluate the coagulopathy.
Tolerance of whole blood transfusion | Day 1, Day 2
  Hemolysis marker rate
Labile blood products transfused in the first 24 hours | 24 hours following hospital admission
  Number of bags administered
Cost of the strategy | Day 30 (or the last day of hospitalization)
  Direct costs of transfusion and the cost of the ICU stay
Biobank establishment | Through study completion, an average of 3 years
  To constitute biobank for biological measurements in research hemorrhagic shock pathophysiology of transfusion resuscitation.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume PELÉE DE SAINT MAURICE, Study Director — Direction Centrale du Service de Santé des Armées (DCSSA); Sylvain AUSSET, Principal Investigator — Institution Nationale des Invalides; Jean-Luc BOSSON, Principal Investigator — Statistical and methodological investigator - Laboratoire TIMC UMR 5525 CNRS Equipe Themas
Locations (6):
- France (6):
  - CHU de La Cavale Blanche - Brest, Brest
  - HIA Percy, Clamart
  - CHU de Grenoble, Grenoble
  - CHU de La Pitié-Salpêtrière, Paris
  - CHU du Kremlin Bicêtre, Paris
  - HIA Sainte Anne, Toulon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spinella PC. Zero preventable deaths after traumatic injury: An achievable goal. J Trauma Acute Care Surg. 2017 Jun;82(6S Suppl 1):S2-S8. doi: 10.1097/TA.0000000000001425. No abstract available. PMID 28333835
- [Background] Bhangu A, Nepogodiev D, Doughty H, Bowley DM. Meta-analysis of plasma to red blood cell ratios and mortality in massive blood transfusions for trauma. Injury. 2013 Dec;44(12):1693-9. doi: 10.1016/j.injury.2012.07.193. Epub 2012 Sep 25. PMID 23021369
- [Background] Johansson PI, Oliveri RS, Ostrowski SR. Hemostatic resuscitation with plasma and platelets in trauma. J Emerg Trauma Shock. 2012 Apr;5(2):120-5. doi: 10.4103/0974-2700.96479. PMID 22787340
- [Background] Cap A, Hunt B. Acute traumatic coagulopathy. Curr Opin Crit Care. 2014 Dec;20(6):638-45. doi: 10.1097/MCC.0000000000000158. PMID 25340382
- [Background] Cap AP, Pidcoke HF, Spinella P, Strandenes G, Borgman MA, Schreiber M, Holcomb J, Tien HC, Beckett AN, Doughty H, Woolley T, Rappold J, Ward K, Reade M, Prat N, Ausset S, Kheirabadi B, Benov A, Griffin EP, Corley JB, Simon CD, Fahie R, Jenkins D, Eastridge BJ, Stockinger Z. Damage Control Resuscitation. Mil Med. 2018 Sep 1;183(suppl_2):36-43. doi: 10.1093/milmed/usy112. PMID 30189070
- [Background] Spahn DR, Bouillon B, Cerny V, Duranteau J, Filipescu D, Hunt BJ, Komadina R, Maegele M, Nardi G, Riddez L, Samama CM, Vincent JL, Rossaint R. The European guideline on management of major bleeding and coagulopathy following trauma: fifth edition. Crit Care. 2019 Mar 27;23(1):98. doi: 10.1186/s13054-019-2347-3. PMID 30917843
- [Background] Godier A, Bacus M, Kipnis E, Tavernier B, Guidat A, Rauch A, Drumez E, Susen S, Garrigue-Huet D. Compliance with evidence-based clinical management guidelines in bleeding trauma patients. Br J Anaesth. 2016 Nov;117(5):592-600. doi: 10.1093/bja/aew317. PMID 27799173
- [Background] Stanworth SJ, Davenport R, Curry N, Seeney F, Eaglestone S, Edwards A, Martin K, Allard S, Woodford M, Lecky FE, Brohi K. Mortality from trauma haemorrhage and opportunities for improvement in transfusion practice. Br J Surg. 2016 Mar;103(4):357-65. doi: 10.1002/bjs.10052. Epub 2016 Feb 3. PMID 26841720
- [Background] Carli P, Pons F, Levraut J, Millet B, Tourtier JP, Ludes B, Lafont A, Riou B. The French emergency medical services after the Paris and Nice terrorist attacks: what have we learnt? Lancet. 2017 Dec 16;390(10113):2735-2738. doi: 10.1016/S0140-6736(17)31590-8. Epub 2017 Jul 25. No abstract available. PMID 28754492
- [Background] Eastridge BJ, Mabry RL, Seguin P, Cantrell J, Tops T, Uribe P, Mallett O, Zubko T, Oetjen-Gerdes L, Rasmussen TE, Butler FK, Kotwal RS, Holcomb JB, Wade C, Champion H, Lawnick M, Moores L, Blackbourne LH. Death on the battlefield (2001-2011): implications for the future of combat casualty care. J Trauma Acute Care Surg. 2012 Dec;73(6 Suppl 5):S431-7. doi: 10.1097/TA.0b013e3182755dcc. PMID 23192066
- [Background] Eastridge BJ, Hardin M, Cantrell J, Oetjen-Gerdes L, Zubko T, Mallak C, Wade CE, Simmons J, Mace J, Mabry R, Bolenbaucher R, Blackbourne LH. Died of wounds on the battlefield: causation and implications for improving combat casualty care. J Trauma. 2011 Jul;71(1 Suppl):S4-8. doi: 10.1097/TA.0b013e318221147b. PMID 21795876
- [Background] Glasgow S, Davenport R, Perkins Z, Tai N, Brohi K. A comprehensive review of blood product use in civilian mass casualty events. J Trauma Acute Care Surg. 2013 Sep;75(3):468-74. doi: 10.1097/TA.0b013e318298efb9. No abstract available. PMID 23928738
- [Background] Doughty H, Glasgow S, Kristoffersen E. Mass casualty events: blood transfusion emergency preparedness across the continuum of care. Transfusion. 2016 Apr;56 Suppl 2:S208-16. doi: 10.1111/trf.13488. PMID 27100758
- [Background] Glasgow SM, Allard S, Rackham R, Doughty H. Going for gold: blood planning for the London 2012 Olympic Games. Transfus Med. 2014 Jun;24(3):145-53. doi: 10.1111/tme.12116. Epub 2014 Apr 18. PMID 24750387
- [Background] Glasgow SM, Allard S, Doughty H, Spreadborough P, Watkins E. Blood and bombs: the demand and use of blood following the London Bombings of 7 July 2005--a retrospective review. Transfus Med. 2012 Aug;22(4):244-50. doi: 10.1111/j.1365-3148.2012.01173.x. PMID 22809430
- [Background] Radwan ZA, Bai Y, Matijevic N, del Junco DJ, McCarthy JJ, Wade CE, Holcomb JB, Cotton BA. An emergency department thawed plasma protocol for severely injured patients. JAMA Surg. 2013 Feb;148(2):170-5. doi: 10.1001/jamasurgery.2013.414. PMID 23426594
- [Background] de Biasi AR, Stansbury LG, Dutton RP, Stein DM, Scalea TM, Hess JR. Blood product use in trauma resuscitation: plasma deficit versus plasma ratio as predictors of mortality in trauma (CME). Transfusion. 2011 Sep;51(9):1925-32. doi: 10.1111/j.1537-2995.2010.03050.x. Epub 2011 Feb 18. PMID 21332727
- [Background] Cardenas JC, Zhang X, Fox EE, Cotton BA, Hess JR, Schreiber MA, Wade CE, Holcomb JB; PROPPR Study Group. Platelet transfusions improve hemostasis and survival in a substudy of the prospective, randomized PROPPR trial. Blood Adv. 2018 Jul 24;2(14):1696-1704. doi: 10.1182/bloodadvances.2018017699. PMID 30030268
- [Background] Holcomb JB, Tilley BC, Baraniuk S, Fox EE, Wade CE, Podbielski JM, del Junco DJ, Brasel KJ, Bulger EM, Callcut RA, Cohen MJ, Cotton BA, Fabian TC, Inaba K, Kerby JD, Muskat P, O'Keeffe T, Rizoli S, Robinson BR, Scalea TM, Schreiber MA, Stein DM, Weinberg JA, Callum JL, Hess JR, Matijevic N, Miller CN, Pittet JF, Hoyt DB, Pearson GD, Leroux B, van Belle G; PROPPR Study Group. Transfusion of plasma, platelets, and red blood cells in a 1:1:1 vs a 1:1:2 ratio and mortality in patients with severe trauma: the PROPPR randomized clinical trial. JAMA. 2015 Feb 3;313(5):471-82. doi: 10.1001/jama.2015.12. PMID 25647203
- [Background] Holcomb JB, del Junco DJ, Fox EE, Wade CE, Cohen MJ, Schreiber MA, Alarcon LH, Bai Y, Brasel KJ, Bulger EM, Cotton BA, Matijevic N, Muskat P, Myers JG, Phelan HA, White CE, Zhang J, Rahbar MH; PROMMTT Study Group. The prospective, observational, multicenter, major trauma transfusion (PROMMTT) study: comparative effectiveness of a time-varying treatment with competing risks. JAMA Surg. 2013 Feb;148(2):127-36. doi: 10.1001/2013.jamasurg.387. PMID 23560283
- [Background] Cap AP, Spinella PC, Borgman MA, Blackbourne LH, Perkins JG. Timing and location of blood product transfusion and outcomes in massively transfused combat casualties. J Trauma Acute Care Surg. 2012 Aug;73(2 Suppl 1):S89-94. doi: 10.1097/TA.0b013e318260625a. PMID 22847102
- [Background] Fox EE, Holcomb JB, Wade CE, Bulger EM, Tilley BC; PROPPR Study Group. Earlier Endpoints are Required for Hemorrhagic Shock Trials Among Severely Injured Patients. Shock. 2017 May;47(5):567-573. doi: 10.1097/SHK.0000000000000788. PMID 28207628
- [Background] Novak DJ, Bai Y, Cooke RK, Marques MB, Fontaine MJ, Gottschall JL, Carey PM, Scanlan RM, Fiebig EW, Shulman IA, Nelson JM, Flax S, Duncan V, Daniel-Johnson JA, Callum JL, Holcomb JB, Fox EE, Baraniuk S, Tilley BC, Schreiber MA, Inaba K, Rizoli S, Podbielski JM, Cotton BA, Hess JR; PROPPR Study Group. Making thawed universal donor plasma available rapidly for massively bleeding trauma patients: experience from the Pragmatic, Randomized Optimal Platelets and Plasma Ratios (PROPPR) trial. Transfusion. 2015 Jun;55(6):1331-9. doi: 10.1111/trf.13098. Epub 2015 Mar 30. PMID 25823522
- [Background] Daban JL, Kerleguer A, Clavier B, Salliol A, Ausset S. [Fresh whole blood transfusion for war surgery: the experience of the Kabul French combat support hospital from 2006 to 2009]. Ann Fr Anesth Reanim. 2012 Nov;31(11):850-6. doi: 10.1016/j.annfar.2012.07.014. Epub 2012 Sep 1. French. PMID 22943967
- [Background] Esnault P, Cungi PJ, Romanat PE, D'Aranda E, Cotte J, Bordes J, Vichard A, Aguillon P, Sailliol A, Meaudre E. [Blood transfusion on battlefield. The Kabul hospital experience]. Ann Fr Anesth Reanim. 2013 Oct;32(10):670-5. doi: 10.1016/j.annfar.2013.06.007. Epub 2013 Aug 13. French. PMID 23953835
- [Background] Ausset S, Meaudre E, Kaiser E, Sailliol A, Hugard L, Jeandel P. [Acute traumatic haemorrhagic shock and transfusion: the French army policy]. Ann Fr Anesth Reanim. 2009 Jul-Aug;28(7-8):707-9. doi: 10.1016/j.annfar.2009.05.011. Epub 2009 Jul 3. No abstract available. French. PMID 19577407
- [Background] McGuigan R, Spinella PC, Beekley A, Sebesta J, Perkins J, Grathwohl K, Azarow K. Pediatric trauma: experience of a combat support hospital in Iraq. J Pediatr Surg. 2007 Jan;42(1):207-10. doi: 10.1016/j.jpedsurg.2006.09.020. PMID 17208567
- [Background] Sailliol A, Clavier B, Cap A, Ausset S. [French European military haemovigilance guidelines]. Transfus Clin Biol. 2010 Dec;17(5-6):315-7. doi: 10.1016/j.tracli.2010.09.001. Epub 2010 Nov 3. French. PMID 21051263
- [Background] Nair PM, Pidcoke HF, Cap AP, Ramasubramanian AK. Effect of cold storage on shear-induced platelet aggregation and clot strength. J Trauma Acute Care Surg. 2014 Sep;77(3 Suppl 2):S88-93. doi: 10.1097/TA.0000000000000327. PMID 25159368
- [Background] Pidcoke HF, Spinella PC, Ramasubramanian AK, Strandenes G, Hervig T, Ness PM, Cap AP. Refrigerated platelets for the treatment of acute bleeding: a review of the literature and reexamination of current standards. Shock. 2014 May;41 Suppl 1:51-3. doi: 10.1097/SHK.0000000000000078. PMID 24662779
- [Background] Nair PM, Pandya SG, Dallo SF, Reddoch KM, Montgomery RK, Pidcoke HF, Cap AP, Ramasubramanian AK. Platelets stored at 4 degrees C contribute to superior clot properties compared to current standard-of-care through fibrin-crosslinking. Br J Haematol. 2017 Jul;178(1):119-129. doi: 10.1111/bjh.14751. Epub 2017 Jun 4. PMID 28580719
- [Background] Bahr MP, Yazer MH, Triulzi DJ, Collins RA. Whole blood for the acutely haemorrhaging civilian trauma patient: a novel idea or rediscovery? Transfus Med. 2016 Dec;26(6):406-414. doi: 10.1111/tme.12329. Epub 2016 Jun 29. PMID 27357229
- [Background] Cotton BA, Podbielski J, Camp E, Welch T, del Junco D, Bai Y, Hobbs R, Scroggins J, Hartwell B, Kozar RA, Wade CE, Holcomb JB; Early Whole Blood Investigators. A randomized controlled pilot trial of modified whole blood versus component therapy in severely injured patients requiring large volume transfusions. Ann Surg. 2013 Oct;258(4):527-32; discussion 532-3. doi: 10.1097/SLA.0b013e3182a4ffa0. PMID 23979267
- [Background] Jenkins D, Stubbs J, Williams S, Berns K, Zielinski M, Strandenes G, Zietlow S. Implementation and execution of civilian remote damage control resuscitation programs. Shock. 2014 May;41 Suppl 1:84-9. doi: 10.1097/SHK.0000000000000133. PMID 24662783
- [Background] Stubbs JR, Zielinski MD, Jenkins D. The state of the science of whole blood: lessons learned at Mayo Clinic. Transfusion. 2016 Apr;56 Suppl 2(Suppl 2):S173-81. doi: 10.1111/trf.13501. PMID 27100754
- [Background] Yazer MH, Jackson B, Sperry JL, Alarcon L, Triulzi DJ, Murdock AD. Initial safety and feasibility of cold-stored uncrossmatched whole blood transfusion in civilian trauma patients. J Trauma Acute Care Surg. 2016 Jul;81(1):21-6. doi: 10.1097/TA.0000000000001100. PMID 27120323
- [Background] Seheult JN, Triulzi DJ, Alarcon LH, Sperry JL, Murdock A, Yazer MH. Measurement of haemolysis markers following transfusion of uncrossmatched, low-titre, group O+ whole blood in civilian trauma patients: initial experience at a level 1 trauma centre. Transfus Med. 2017 Feb;27(1):30-35. doi: 10.1111/tme.12372. Epub 2016 Oct 12. PMID 27730689
- [Background] Savage SA, Zarzaur BL, Pohlman TH, Brewer BL, Magnotti LJ, Croce MA, Lim GH, Martin AC. Clot dynamics and mortality: The MA-R ratio. J Trauma Acute Care Surg. 2017 Oct;83(4):628-634. doi: 10.1097/TA.0000000000001637. PMID 28930957
- [Background] Einersen PM, Moore EE, Chapman MP, Moore HB, Gonzalez E, Silliman CC, Banerjee A, Sauaia A. Rapid thrombelastography thresholds for goal-directed resuscitation of patients at risk for massive transfusion. J Trauma Acute Care Surg. 2017 Jan;82(1):114-119. doi: 10.1097/TA.0000000000001270. PMID 27805995
- [Background] Gonzalez E, Moore EE, Moore HB, Chapman MP, Chin TL, Ghasabyan A, Wohlauer MV, Barnett CC, Bensard DD, Biffl WL, Burlew CC, Johnson JL, Pieracci FM, Jurkovich GJ, Banerjee A, Silliman CC, Sauaia A. Goal-directed Hemostatic Resuscitation of Trauma-induced Coagulopathy: A Pragmatic Randomized Clinical Trial Comparing a Viscoelastic Assay to Conventional Coagulation Assays. Ann Surg. 2016 Jun;263(6):1051-9. doi: 10.1097/SLA.0000000000001608. PMID 26720428
- [Background] Zatta AJ, McQuilten ZK, Mitra B, Roxby DJ, Sinha R, Whitehead S, Dunkley S, Kelleher S, Hurn C, Cameron PA, Isbister JP, Wood EM, Phillips LE; Massive Transfusion Registry Steering Committee. Elucidating the clinical characteristics of patients captured using different definitions of massive transfusion. Vox Sang. 2014 Jul;107(1):60-70. doi: 10.1111/vox.12121. Epub 2014 Apr 2. PMID 24697251
- [Background] Godier A, Samama CM, Susen S. [Management of massive bleeding in 2013: seven questions and answers]. Transfus Clin Biol. 2013 May;20(2):55-8. doi: 10.1016/j.tracli.2013.02.015. Epub 2013 Apr 12. French. PMID 23587620
- [Background] Hamada SR, Rosa A, Gauss T, Desclefs JP, Raux M, Harrois A, Follin A, Cook F, Boutonnet M; Traumabase(R) Group; Attias A, Ausset S, Boutonnet M, Dhonneur G, Duranteau J, Langeron O, Paugam-Burtz C, Pirracchio R, de St Maurice G, Vigue B, Rouquette A, Duranteau J. Development and validation of a pre-hospital "Red Flag" alert for activation of intra-hospital haemorrhage control response in blunt trauma. Crit Care. 2018 May 5;22(1):113. doi: 10.1186/s13054-018-2026-9. PMID 29728151
- [Background] Nunez TC, Voskresensky IV, Dossett LA, Shinall R, Dutton WD, Cotton BA. Early prediction of massive transfusion in trauma: simple as ABC (assessment of blood consumption)? J Trauma. 2009 Feb;66(2):346-52. doi: 10.1097/TA.0b013e3181961c35. PMID 19204506
- [Background] Pommerening MJ, Goodman MD, Holcomb JB, Wade CE, Fox EE, Del Junco DJ, Brasel KJ, Bulger EM, Cohen MJ, Alarcon LH, Schreiber MA, Myers JG, Phelan HA, Muskat P, Rahbar M, Cotton BA; MPH on behalf of the PROMMTT Study Group. Clinical gestalt and the prediction of massive transfusion after trauma. Injury. 2015 May;46(5):807-13. doi: 10.1016/j.injury.2014.12.026. Epub 2015 Feb 4. PMID 25682314
- [Background] Yazer MH, Delaney M, Doughty H, Dunbar NM, Al-Riyami AZ, Triulzi DJ, Watchko JF, Wood EM, Yahalom V, Emery SP. It is time to reconsider the risks of transfusing RhD negative females of childbearing potential with RhD positive red blood cells in bleeding emergencies. Transfusion. 2019 Dec;59(12):3794-3799. doi: 10.1111/trf.15569. Epub 2019 Oct 18. No abstract available. PMID 31625172
- [Background] Martinaud C, Civadier C, Ausset S, Verret C, Deshayes AV, Sailliol A. In vitro hemostatic properties of French lyophilized plasma. Anesthesiology. 2012 Aug;117(2):339-46. doi: 10.1097/ALN.0b013e3182608cdd. PMID 22739764
- [Background] Raux M, Le Manach Y, Gauss T, Baumgarten R, Hamada S, Harrois A, Riou B, Duranteau J, Langeron O, Mantz J, Paugam-Burtz C, Vigue B; TRAUMABASE Group. Comparison of the Prognostic Significance of Initial Blood Lactate and Base Deficit in Trauma Patients. Anesthesiology. 2017 Mar;126(3):522-533. doi: 10.1097/ALN.0000000000001490. PMID 28059838
- [Background] Regnier MA, Raux M, Le Manach Y, Asencio Y, Gaillard J, Devilliers C, Langeron O, Riou B. Prognostic significance of blood lactate and lactate clearance in trauma patients. Anesthesiology. 2012 Dec;117(6):1276-88. doi: 10.1097/ALN.0b013e318273349d. PMID 23168430
- [Background] Manikis P, Jankowski S, Zhang H, Kahn RJ, Vincent JL. Correlation of serial blood lactate levels to organ failure and mortality after trauma. Am J Emerg Med. 1995 Nov;13(6):619-22. doi: 10.1016/0735-6757(95)90043-8. PMID 7575797
- [Background] Abramson D, Scalea TM, Hitchcock R, Trooskin SZ, Henry SM, Greenspan J. Lactate clearance and survival following injury. J Trauma. 1993 Oct;35(4):584-8; discussion 588-9. doi: 10.1097/00005373-199310000-00014. PMID 8411283
- [Background] Smith IM, Crombie N, Bishop JR, McLaughlin A, Naumann DN, Herbert M, Hancox JM, Slinn G, Ives N, Grant M, Perkins GD, Doughty H, Midwinter MJ; RePHILL Trial Collaborators. RePHILL: protocol for a randomised controlled trial of pre-hospital blood product resuscitation for trauma. Transfus Med. 2018 Oct;28(5):346-356. doi: 10.1111/tme.12486. Epub 2017 Nov 28. PMID 29193548
- [Background] Boutonnet M, Abback P, Le Sache F, Harrois A, Follin A, Imbert N, Cap AP, Trichereau J, Ausset S; Traumabase Group. Tranexamic acid in severe trauma patients managed in a mature trauma care system. J Trauma Acute Care Surg. 2018 Jun;84(6S Suppl 1):S54-S62. doi: 10.1097/TA.0000000000001880. PMID 29538226
- [Background] Riou B, Thicoïpe M, Atain-Kouadio P, Carli P. Comment evaluer la gravité? In: France S de, editor. Actualités en réanimation préhospitalière, Paris: Société française d'éditions médicales; 2002.
- [Background] Duranteau J, Asehnoune K, Pierre S, Ozier Y, Leone M, Lefrant J-Y. Recommandations sur la réanimation du choc hémorragique. Anesthésie & Réanimation 2015;1:62-74. https://doi.org/10.1016/j.anrea.2014.12.007.
- [Background] Massive transfusion in trauma guidelines. American College of Surgeons. Quality improvement project: trauma resuscitation best practice guidelines. Chicago (IL): American College of Surgeons 2013.
- [Background] Miller RD. Massive blood transfusions: the impact of Vietnam military data on modern civilian transfusion medicine. Anesthesiology. 2009 Jun;110(6):1412-6. doi: 10.1097/ALN.0b013e3181a1fd54. PMID 19417598
- [Background] Brohi K, Levy H, Boffard K, Riou B, Kiepert P, Zielske D. Normalization of lactate within 8 hours or ≥20% clearance in initial 2 hours correlates with outcomes from traumatic hemorrhagic shock. Critical Care Medicine 2011;39:177.
- [Derived] Brunskill SJ, Disegna A, Wong H, Fabes J, Desborough MJ, Doree C, Davenport R, Curry N, Stanworth SJ. Blood transfusion strategies for major bleeding in trauma. Cochrane Database Syst Rev. 2025 Apr 24;4(4):CD012635. doi: 10.1002/14651858.CD012635.pub2. PMID 40271704